CLINICAL TRIAL: NCT03753503
Title: Physical Training Induced Plasticity of Motor Control Mechanisms in Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Wroclaw Medical University (Other); University School of Physical Education, Krakow, Poland (Other)
Responsible Party: Principal Investigator, Jaroslaw Marusiak, Principal Investigator, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0247/p01/2010/70
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease; Physical Activity
Keywords: Parkinson's disease; intensive interval training; motor function; executive function; neuroplasticity
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PD-TR (Experimental): Intervention:
  exercise, dose: 8-week HIIT program (three times a week) & conventional physical therapy
  Interventions: Behavioral: exercise; Behavioral: conventional physical therapy
- PD-NTR (Active Comparator): conventional physical therapy
  Interventions: Behavioral: conventional physical therapy
- Healthy controls (No Intervention): healthy controls without any kind of therapy

INTERVENTIONS:
Behavioral: exercise — exercised three times a week in the 8-week HIIT program
  Arms: PD-TR
Behavioral: conventional physical therapy
  Arms: PD-NTR; PD-TR

SUMMARY:
There are experimental evidences of the important role of exercise in the PD, that induces similar effects to pharmacotherapy. So far, the mechanisms of the impact of these changes on the brain subcortical and cortical regions functioning, motor activities and cognitive functions are still not clear. The aim of this longitudinal human experiment is to examine the effects of cycle of 8-week high-intensity interval training (HIIT) on: (i) neurophysiological function of cortical motor structures and skeletal muscle actvity, (ii) psychomotor behavior critically associated with dopamine dependent neural structures functioning and (iii) neurotrophic factors' secretion level in blood. The investigators will recruit 40 PD individuals, who will be divided into two groups: one of them will perform two 8-weeks cycle of HIIT (PD-TR), and the other will not (PD-NTR). The investigators will recruit also 20 age-matched healthy controls (H-CO) as additional control group who will not perform the HIIT. All PD subjects will be examined during their medication "OFF-phase" pre HIIT and 1 week-, 1 month-POST cycle of HIIT. The subject from H-CO will be tested only once. To examine the assumed HIIT-induced changes in brain functioning the investigators will use: (i) EEG (recorded simultaneously with EMG) methods to assess an amplitude, location and directionality of brain electrical current of cortical regions and strength of intra-cortical network interactions during motor tasks performance. During the EEG experiments the subjects will perform (i) bimanual anti-phase DA level dependent motor tasks (during which the investigators will record EMG, force). The investigators will also assess motor and non-motor symptoms of PD and functional test of manual dexterity to evaluate a quality psychomotor behavior.

Using these methods the investigators will determine in detail the mechanisms of functioning of the CNS in PD patients, with emphasis on the cortical interactions that are dependent on synthesis and DA transmission. The results of the study will help to answer the fundamental questions about HIIT induced neuroplasticity in PD patients, as well as complement the lack in knowledge about the mechanisms of exercise-induced changes in PD, and as a consequence it could enrich the golden standard of treatment in PD from pharmacotherapy toward implementation of precise evidence based rehabilitation.

DETAILED DESCRIPTION:
I. Research Project Objectives

Aim 1. To characterize an influence of 8-week HIIT cycle on neurophysiological functions (NPFs) of: (i) motor cortical structures, (that are critically dependant on the presynaptic DA availability), using EEG, and (ii) skeletal muscles engaged in motor task, using surface EMG. The following neurophysiological functions of CNS will be tested during performance of the DA availability-dependant self initiated bimanual motor tasks: (i) a level of activation of cortical structures, and (ii) strength of functional coupling between neural structures. For skeletal muscles NPFs', the investigators will study a strategy of motor units activation. Also, since the investigators will record EEG and EMG simultaneously, the investigators will assess strength of cortico-muscular coupling.

Hypothesis 1. NPFs will improve after the 8-week HIIT cycle compared to baseline in the PD-TR group, and will sustain one month post HIIT. Namely, the investigators speculate that for the motor in CNS activity, it will be: (1) primary motor cortex (M1), supplementary motor area (SMA); (2) decrease of activation of lateral premotor cortex (PMC) and cerebellum; with simultaneous (3) increase of functional coupling of: dorsolateral prefrontal cortex (DLPFC) with M1, PMC, SMA and cerebellum; (4) decrease of functional coupling between M1, PMC, SMA, cerebellum and parietal cortex. For the skeletal muscle function it will be an improvement in recruitment strategy of motor units. Taking into the data from the simultaneous recording of electrical activity of brain cortex and skeletal muscles engaged in motor tasks, the investigators assume strengthening of corticomuscular coupling. In the PD-NTR group NPFs will not improve or even will be worsened in the same time interval.

Aim 2. To characterize an influence of the 8-week HIIT cycle on the psychomotor behaviors (PMBs), critically dependant on the DA availability and brain's NPFs. The following PMBs will be tested during several experiments: (1) self initiated bimanual anti-phase movement tasks during the simultaneous EEG, EMG and force recordings (2) all motor and non-motor PD symptoms evaluation, based on neurological assessment, (3) overall cognitive function and specifically aspects of executive function using psychological tests.

Hypothesis 2. PMBs will improve after the 8-week HIIT cycle compared to baseline in the PD-TR group, and will sustain one month post HIIT, as a consequence of the improvements of presynaptic striatal DA availability and NPFs, The PMBs improvement will not be present in the PD-NTR group, or even the PMBs will be worsened in the same time interval.

Aim 3. To evaluate: (i) the effect of the 8-week HIIT cycle on BDNF, NGF, IGF-1 secretion level in blood treated as markers of neuroplasticity efficiency (expressed in exercise-induced increase of presynaptic DA level, and improvement of NPF' and PMBs).

Hypothesis 3. The secretion level of the BDNF, NGF and IGF-1 will increase after the first and second bout of HIIT cycle compared to baseline in the PD-TR group, and will sustain one month post HIIT. In contrary to PD-TR group, the improvement in BDNF, NGF and IGF-1 secretion level will not be present in the PD-NTR group or even their level will decrease.

II. Justification for tackling specific scientific problems by the proposed project.

II.1. EEG and EMG application to evaluate NPFs of brain cortical structures and skeletal muscles II.1.1. A level of activation of neural cortical structures will be evaluated with EEG averaging and source analysis (cortical neurons circuits).

II.1.2. Strength of functional coupling between the neural cortical structures will be assessed with EEG-EEG coherence analysis:

II.1.3. Motor units activation strategy of skeletal muscle engaged during motor task will be tested with surface EMG standard analysis and SSA.

II.1.4. Strength of functional cortico-muscular coupling will be evaluated with analysis of coherence between EEG and EMG signals:

II.2. PMBs will be evaluated based on motor and cognitive tasks performance, and neurological and psychological tests/scales:

II.2.1. Self initiated bimanual anti-phase index finger movements and bimanual dexterity tasks will be assessed during simultaneous EEG, EMG and force recordings based on analysis of force development, respectively.

II.2.2. Motor and non-motor PD symptoms evaluation, based on neurological assessment using the whole Unified Parkinson's Disease Rating Scale (UPDRS) and Hoehn and Yahr scale (H&Y). Also, for the purpose of correlation estimation between the bimanual dexterity function described in points II.2.1 the investigators will choose from the UPDRS the scores dedicated for manual and bimanual function. Namely, the investigators will analyze parkinsonian bradykinesia scores of the affected/more affected upper extremity based on the items 23-25 from UPDRS (finger tapps, opening and closing hands, pronation-supination hands movement; respectively). The investigators will also analyze: (i) a performance of daily life manual functions based on the items 8-11 from UPDRS (handwriting, cutting food and handling utensils, dressing, hygiene; respectively). Additionally, the investigators will assess the quality of life using Schwab and England Daily Living Activity Scale (S&E DLA) (Fahn and Elton, 1987).

II.2.3. Psychological assessment of executive function using two tests: the Trail Making Test (TMT) and Stroop Test (ST). In both the TMT and ST tests the time taken to complete the test is used as the performance measure with shorter time as better performance. Also, to exclude the patients with dementia the investigators will apply Mini Mental State Examination test (MMSE) (Folstein et al., 1975).

II.3. Neurotrophic factors secretion in blood By using the enzyme-linked immunosorbent assay (ELISA technique), the investigators will assess secretion of serum BDNF, NGF, IGF-1 in blood, that are responsible for neurogenesis, synaptogenesis, angiogenesis.

III. Work plan The project realization is scheduled for 24 months. The project will enroll two PD patients' groups: PD-TR - the PD patients who will perform physical training cycle; PD-NTR - non-trained PD patients and one H-CO - healthy control group that will not perform the HIIT cycles.

The project will start with baseline testing session (PRE-HIT) in the both PD groups. Then the PD-TR group will perform the 8-week HIIT cycle, and the PD-NTR group will not perform HIIT cycle in this time period. Then, 1 week-, and one month post HIIT cycle cessation the investigators will perform testing sessions in the PD-TR and PD-NTR group. The healthy control group will be tested only in one time point, when the lab space will not be occupied with PD patients tests.

IV. Research methodology

IV.1. Research design This project will be a longitudinal, randomized (opaque envelopes randomization) controlled study with 3 arms. The investigators will recruit 40 PD individuals, who will be randomly allocated into two equal groups: PD-TR (N=20) and PD-NTR (N=20). The investigators will compare the results from these two groups to explore a longitudinal effect HIIT cycles on measurement outcomes. Additionally, the investigators will recruit a healthy control group (H-CO; N=20) that will be tested only once, and will constitute "healthy state" condition for comparisons with both PD patients groups. The comparison of PD-NTR with H-CO will show us the mechanisms of pathological changes in PD patients and comparison of PD-TR with H-CO will give us an opportunity to explore the character of mechanisms (restoration or compensation) of HIIT induced changes in PD patients.

The 40 PD individuals, will be qualified to our study after being diagnosed to have an idiopatic PD, based on neurological assessment. The diagnosis of Parkinson's disease will be based on medical history, physical and neurological examinations and response to L-dopa. IV.2.2. Subjects recruitment. The PD subjects will be recruited from Neurology Clinic, Wroclaw Medical University (WMU) in Wroclaw, Poland, where the person performing the neurological PD patients evaluation in our project (Budrewicz Slawomir, M.D, Ph.D.) is employed as movement disorders neurologists and consult PD patients there. Taking into account the capabilities and top position of the WMU, the investigators are sure that the investigators are able to recruit and finally qualify 40 PD patients. The healthy elderly control group of subjects will be recruited based on: (i) public advertisement and (ii) contacts with the Universities of the Third Age and the Seniors' Clubs around the Warsaw city.

IV.2. Training procedures The patients from PD-TR group will perform 8-week HIIT cycle. The 8-week HIIT program will consist of three weekly 1-hour training sessions (each consisting of a 10-min warm-up, 40 min of high-intensity interval exercise and a 10-min cool-down phase at a slow voluntary speed) performed on a stationary cycle ergometer (MONARK, Ergomedic 874E, Sweden) that will measure cadence (revolutions per minute; [rpm]) and power [W]. During each training session, the interval exercise will consist of 8 sets of 5-min intervals, including 3 min of cycling at ≥ 60 [rpm] but preferably at 80-90 [rpm] (fast phase of interval) and 2 min of cycling at ≤ 60 [rpm] (slow phase of interval). The patients in the PD-TR group will be rhythmically cued by a metronome and verbally encouraged by an instructor to pedal with the set speed appropriate for the fast and slow phases. The cadence values will be presented to each subject in real time on a screen as feedback to control the rpm during the different interval phases. The heart rate (HR; beats per minute [bpm]) measured using a Polar system (Polar, Finland), cadence [rpm], and power [W] will be monitored and collected during each training session. Training supervisor will adjust the resistance for each patient to ensure cycling at each patient's target heart rate (THR) and with appropriate speed. PD patients will cycle at 60%-75% of their individualized HRmax (maximal heart rate). The PD patients will be encouraged to cycle faster (80-90 rpm or 30% faster than their voluntary pedaling rate) during the fast phase of interval and to increase his/her THR every 2 weeks by 5% (60% of the HRmax during 1-2 week, 65% during 3-4 week, 70% during 5-6 week, and 75% during 7-8 week of training period). Additionally, the patients' perceptions of the exercise intensity (for the fast and slow phases of the interval) will be assessed using the Borg Rating of Perceived Exertion (RPE) (Borg, 1982).

IV.3. Measurement procedures All PD subjects will be examined during their medication off-phase, i.e. after an overnight 12-hours withdrawal of anti-parkinsonian drugs (24-hours for extended release medications). The testing sessions' sequence for specific methods is as follows: 1'st day - (i) blood sampling; (ii) psychological, neurological and functional tests -> 2'nd day - (i) EEG + EMG + force.

IV.4. Statistical analysis The investigators will first perform a between-group comparison for all demographics and clinical characteristics to check for baseline differences. This will be done using the two-tailed Student's t test or Mann-Whitney U tests for normally and non-normally distributed data or the Fisher's exact test for contingency data. Repeated measures analysis of variance will be used to perform a between-group comparison of changes in the testing points. Significant main effects will then be subjected to a post-hoc pair-wise comparison primarily between PD-TR and PD-NTR, and PD-TR and H-CO. Correlation analysis (Pearson or Spearman correlation coefficient) will be performed between EEG, EMG (describing NPFs), PMBs, and neuroplasticity markers outcomes. For all analyses, a significance level will be set to α=0.05 with Bonferroni adjustments for multiple comparisons when necessary.

ELIGIBILITY:
Inclusion Criteria:

* for PD patients: age 55-75 years-old; diagnosis of idiopathic PD; and modified Hoehn and Yahr stages between 1.5 and 3
* for healthy controls: lack of neurological disorders

Exclusion Criteria:

* for PD patients: (i) presence of other neurological disorders, (2) any cardiovascular and respiratory system restrictions and/or motor deficits that could limit performance in high-speed pedaling on a cycle ergometer or in the conventional physical therapy and (3) practicing any regular physical activity except for physical therapy for PD
* for healthy controls: presence of neurological disorders

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2015-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Electroencephalography (EEG) - electrical activity of brain cortex recorded from scalp using surface electrodes. | Baseline
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 64-chanel system. The recordings will be conducted during bimanual motor tasks and at rest. The recordings will be expressed in microvolts [µV].
Electroencephalography (EEG) - electrical activity of brain cortex recorded from scalp using surface electrodes. | 1-week-post HIIT cycle
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 64-chanel system. The recordings will be conducted during bimanual motor tasks and at rest. The recordings will be expressed in microvolts [µV].
Electroencephalography (EEG) - electrical activity of brain cortex recorded from scalp using surface electrodes. | 1-month-post HIIT cycle
  To evaluate neurophysiological functions of brain cortical structures, electroencephalography (EEG - electrical activity of brain cortex) will be recorded from scalp using 64-chanel system. The recordings will be conducted during bimanual motor tasks and at rest. The recordings will be expressed in microvolts [µV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | Baseline
  To evaluate neurophysiological functions of muscles engaged in an activity (hand and forearm muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during bimanual motor tasks and at rest. The recordings will be expressed in milivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1-week-post HIIT cycle
  To evaluate neurophysiological functions of muscles engaged in an activity (hand and forearm muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during bimanual motor tasks and at rest. The recordings will be expressed in milivolts [mV].
Electromyography (EMG) - recordings of electrical activity of skeletal muscles using surface electrodes. | 1-month-post HIIT cycle
  To evaluate neurophysiological functions of muscles engaged in an activity (hand and forearm muscles), electromyography (EMG - recordings of electrical activity of skeletal muscles) will be collected using surface electrodes, during bimanual motor tasks and at rest. The recordings will be expressed in milivolts [mV].
BDNF - brain derived neurotrophic factor | Baseline
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1-week-post HIIT cycle
  BDNF secretion level in blood expressed in [pg/mL]
BDNF - brain derived neurotrophic factor | 1-month-post HIIT cycle
  BDNF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | Baseline
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1-week-post HIIT cycle
  NGF secretion level in blood expressed in [pg/mL]
NGF - nerve growth factor | 1-month-post HIIT cycle
  NGF secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | Baseline
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1-week-post HIIT cycle
  IGF 1 secretion level in blood expressed in [pg/mL]
IGF 1 - insulin-like growth factor 1 | 1-month-post HIIT cycle
  IGF 1 secretion level in blood expressed in [pg/mL]
Force measurements of both hands' index fingers motor control | Baseline
  force development measurements of self initiated bimanual anti-phase index finger movements, using force transducers system. The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
Force measurements of both hands' index fingers motor control | 1-week-post HIIT cycle
  force development measurements of self initiated bimanual anti-phase index finger movements, using force transducers system. The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
Force measurements of both hands' index fingers motor control | 1-month-post HIIT cycle
  force development measurements of self initiated bimanual anti-phase index finger movements, using force transducers system. The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
Force measurements of bimanual dexterity function | Baseline
  force development measurements of self initiated bimanual anti-phase hand grip-load function, using force transducers system. The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
Force measurements of bimanual dexterity function | 1-week-post HIIT cycle
  force development measurements of self initiated bimanual anti-phase hand grip-load function, using force transducers system.The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
Force measurements of bimanual dexterity function | 1-month-post HIIT cycle
  force development measurements of self initiated bimanual anti-phase hand grip-load function, using force transducers system. The force will be expressed in [N], the time of force development in [s] and the rate of force development in [N/s].
TMT-A - trail making test, part A | Baseline
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1-week-post HIIT cycle
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-A - trail making test, part A | 1-month-post HIIT cycle
  TMT-A is a psychological measure of cognitive processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | Baseline
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1-week-post HIIT cycle
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
TMT-B - trail making test, part B | 1-month-post HIIT cycle
  TMT-B is a psychological measure of executive function, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | Baseline
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1-week-post HIIT cycle
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-I - Stroop Test, part I | 1-month-post HIIT cycle
  ST-I is used as a psychological measure of processing speed, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | Baseline
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1-week-post HIIT cycle
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].
ST-II - Stroop Test, part II | 1-month-post HIIT cycle
  ST-II is used as a psychological measure of selective attention and inhibition, measured as performance time (the shorter the time the better performance), expressed in [s].

SECONDARY OUTCOMES:
UPDRS - unified Parkinson's disease rating scale | Baseline
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1-week-post HIIT cycle
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
UPDRS - unified Parkinson's disease rating scale | 1-month-post HIIT cycle
  Motor and non-motor Parkinson's disease signs/symptoms will be evaluated using UPDRS (sections I - III, that include the items 1 -31). Each item is expressed in [points] from 0 to 4 points, with an interpretation that the higher value means the severe accentuation of sign/symptom. The total score will be reported, as the sum of the points of the sections I-III (the score in the range 0 - 176 points) and each section's score will be reported as well, i.e.: the sum of the points of the section I (sum of points for items 1-4 in the range 0 - 16 points), the sum of the points of the section II (sum of points for items 5-17 in the range 0 - 52 points), the sum of the points of the section III (sum of points for items 18-31 in the range 0 - 108 points).
H&Y scale - Hoehn and Yahr scale | Baseline
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1-week-post HIIT cycle
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
H&Y scale - Hoehn and Yahr scale | 1-month-post HIIT cycle
  Parkinson's disease stage evaluation using H&Y scale, expressed in [points] from 1 to 5 points. The modified version of the H&Y scale will be used, in which: the score 1 means - unilateral involvement only; the score 1.5 means - unilateral and axial involvement; the score 2 means - bilateral involvement without impairment of balance; the score 2.5 means - mild bilateral disease with recovery on pull test; the score 3 means - mild to moderate bilateral disease, some postural instability, physically independent; the score 4 means - severe disability, still able to walk or stand unassisted; the score 5 means - wheelchair bound or bedridden unless aided.
S&E DLA scale - Schwab and England Daily Living Activity Scale | Baseline
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score decribes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1-week-post HIIT cycle
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score decribes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
S&E DLA scale - Schwab and England Daily Living Activity Scale | 1-month-post HIIT cycle
  S&E DLA scale measure of daily function of Parkinson's disease patients, expressed in [%] from 100 to 0 % (with the higher % value as the better score). The 100% score means that the person is completely independent; able to do all chores without slowness, difficulty or impairment; essentially normal; unaware of any difficulty. The 0% score decribes the person bedridden with the only vegetative functions such as swallowing; bladder and bowel functions are not functioning.
MMSE - Mini Mental State Examination | Baseline
  MMSE will be used to to exclude the Parkinson's disease patients with cognitive impairment, expressed in [points]in the range from 0 to 30 points. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. A score of 23 or lower is indicative of cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jarosław Marusiak, PhD, Principal Investigator — Wroclaw University of Health and Sport Sciences

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Marusiak J, Zeligowska E, Mencel J, Kisiel-Sajewicz K, Majerczak J, Zoladz JA, Jaskolski A, Jaskolska A. Interval training-induced alleviation of rigidity and hypertonia in patients with Parkinson's disease is accompanied by increased basal serum brain-derived neurotrophic factor. J Rehabil Med. 2015 Apr;47(4):372-5. doi: 10.2340/16501977-1931. PMID 25510618
- [Result] Zoladz JA, Majerczak J, Zeligowska E, Mencel J, Jaskolski A, Jaskolska A, Marusiak J. Moderate-intensity interval training increases serum brain-derived neurotrophic factor level and decreases inflammation in Parkinson's disease patients. J Physiol Pharmacol. 2014 Jun;65(3):441-8. PMID 24930517
- See also: The New York Times article about our findings. Author: Jane E. Brody; Title: Why Your Workout Should Be High-Intensity, autorka: JANE E. BRODY — https://well.blogs.nytimes.com/2015/01/26/sweaty-answer-to-chronic-illness/?_r=1